CLINICAL TRIAL: NCT05663099
Title: Cauterization of the Anterior Ethmoidal Artery by Transconjunctival Approach
Acronym: AEA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8719
Record Dates: First submitted 2022-12-14; First posted 2022-12-23 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2022-12

CONDITIONS: Epistaxis, Anterior Ethmoid Artery
Keywords: Epistaxis; Anterior Ethmoid Artery; Arterial hypertension; Hemostasis disorders; Endoscopic sphenopalatine artery; Endonasal endoscopic; Anterior ethmoidectomy
MeSH Terms: conditions — Epistaxis; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The incidence of epistaxis varies from 7 to 14% in the general population and represents 30 per 100,000 emergency room admissions in adults. Most nasal bleeding is self-limiting without the need for specific medical treatment. Cauterization under local anesthesia and control of medical comorbidities (arterial hypertension and hemostasis disorders) are effective in most cases. In case of failure of cauterization or in case of more posterior epistaxis, an antero-posterior packing can be put in place for 48 hours. In case of failure or recurrence of packing removal, endoscopic sphenopalatine artery (SPA) ligation or embolization is proposed. In case of persistent epistaxis despite hemostasis of the PSA, ligation of the anterior ethmoidal artery (AEA) is recommended. This artery cannot be embolized because of the risk to the ophthalmic artery. The ligation of the AEA is most often performed via the external paracanthal approach. It can also be performed by endonasal endoscopic approach but involves the performance of an anterior ethmoidectomy, a long surgery with a significant risk of complications. Its identification by the endonasal route is complicated in the event of abundant bleeding. Moreover, its endoscopic cauterization is difficult if the artery is not procidente. The transconjunctival approach avoids a visible scar and the complications of an ethmoidectomy.

DETAILED DESCRIPTION:
The objective of the study was to compare the efficacy of transconjunctival and external cauterization of the anterior ethmoidal artery in patients with refractory epistaxis

ELIGIBILITY:
Inclusion criteria:

* Male or female (age ≥18 years)
* Persistent epistaxis after meching
* Having required transconjunctival anterior ethmoidal artery cauterization surgery
* Subject operated at the University Hospitals of Strasbourg between 01/01/2015 and 01/05/2023
* Subject not objecting to the reuse of his/her data for scientific research purposes.

Exclusion Criteria:

- Subject who has expressed opposition to the reuse of his/her data for scientific research purposes.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient having un persistent epistaxis after meching
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02-07 (Estimated)

PRIMARY OUTCOMES:
To retrospectively compare the efficacy of transconjunctival and external cauterization of the anterior ethmoidal artery in patients with refractory epistaxis | Files analysed retrospectively from January 01, 2015 to May 01, 2023 will be examined
  The endpoint is the efficacy of the technique with the presence of postoperative epistaxis recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'ORL et de Chirurgie Cervico-Faciale - CHU de Strasbourg - France, Strasbourg, France